CLINICAL TRIAL: NCT06085755
Title: Ph 1/2 Study of Trastuzumab Deruxtecan(T-DXd) and Afatinib Combination in HER2-low Advanced Gastric Cancer(VIKTORY-2)
Brief Title: Trastuzumab Deruxtecan(T-DXd) and Afatinib Combination in HER2-low Advanced Gastric Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jeeyun Lee (Other)
Responsible Party: Sponsor-Investigator, Jeeyun Lee, Principal Investigator, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-09-015
Record Dates: First submitted 2023-09-10; First posted 2023-10-17 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Stomach Neoplasm
MeSH Terms: conditions — Stomach Neoplasms | interventions — trastuzumab deruxtecan; Afatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trastuzumab deruxtecan + Afatinib (Experimental): The first part (PART A) will be in combination with T-DXd the starting dose of 20 mg afatinib MWF will be escalated to reach a maximum tolerated dose in patients with advanced gastric cancer patients with HER2-low, as defined by dose-limiting toxicity.
  The second part (PART B) will be expansion cohort, in which Afatinib will be taken in combination with T-DXd according to the recommended Phase 2 dose(RP2D) confirmed through Part A from cycle 1.
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Afatinib

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — Trastuzumab deruxtecan will be administered 6.4mg/kg or 5.4mg/kg iv infusion q 3weeks as one cycle.
  Other Names: T-DXd
Drug: Afatinib — Afatinib will be administered orally 20mg ~40mg once a day or three times a week(Monday, Wednesday, Friday [MWF]) or twice weekly (Monday, Thursday [MT]) for 3weeks as one cycle.
  Other Names: Giotrif

SUMMARY:
Despite recent advances, the prognosis of patients with advanced gastric cancer remains poor. At present, regimens that combine a platinum and fluorouracil agent either alone or in combination with a third drug such as epirubicin or taxane constitute the most effective treatment option in the first-line metastatic setting, resulting in a median OS of approximately 10 months. In the second-line setting, ramucirumab (a vascular endothelial growth factor receptor 2 antagonist) was recently approved by the United States Food and Drug Administration, and has demonstrated modest activity in patients with advanced gastric or GEJ adenocarcinoma who progressed after first-line platinum- or fluoropyrimidine-containing chemotherapy. Median OS was 5.2 months in the ramucirumab group versus 3.8 months in the placebo group.

At the updated DCO of 03 June 2020 in the DS8201-A-J202 (DESTINY-Gastric01) study in HER2-positive GC or GEJ adenocarcinoma subjects assigned to T-DXd 6.4 mg/kg, T-DXd further demonstrated clinically meaningful efficacy. The median OS was 12.5 months for the T-DXd group and 8.9 months for the physician's choice group (HR = 0.60, 95% CI: 0.42, 0.86). In a prespecified subgroup analysis, the percentages of patients with an objective response were analyzed in HER2-low group. The response rate in HER2 2+ was 29% (8 of 28) with T-DXd monotherapy.

Refer to the figure below for the response rate in HER2-low group in previous DESTINY trials.

This is a two part, phase I/Ⅱ, open-label, single center study of afatinib in combination with T-DXd, in 2L/3L gastric cancer patients with HER2-low. The study design allows an investigation of combination dose of afatinib with T-DXd, with intensive safety monitoring to ensure the safety of the patients.

DETAILED DESCRIPTION:
Patients who 2nd and 3rd line and expected propositions with histologically confirmed metastatic and/or recurrent gastric adenocarcinoma, an Eastern Cooperative Oncology Group performance status of 0 or 1, and at least one measurable lesion according to the RECIST 1.1 are eligible. Adequate hematologic function, hepatic function, and renal function are required. Patients with other concurrent uncontrolled medical diseases and/or other tumors are also excluded.

The first part (PART A) will be in combination with T-DXd the starting dose of 20 mg afatinib MWF will be escalated to reach a maximum tolerated dose in patients with advanced gastric cancer patients with HER2-low, as defined by dose-limiting toxicity.

The second part (PART B) will be expansion cohort, in which Afatinib will be taken in combination with T-DXd according to the recommended Phase 2 dose(RP2D) confirmed through Part A from cycle 1. PK samples will be collected at designated points, in both Part A and Part B.

Tumor evaluation using modified RECIST 1.1 will be conducted at screening (within 28 days prior to first dose) and every 6 weeks relative to the date of first dose, up to week 40, then every 12 weeks until objective disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of fully informed consent prior to any study specific procedures.
2. Patients must be ≥ 19 years of age
3. Has a pathologically documented advanced or metastatic adenocarcinoma of gastric or gastroesophageal junction with at least one measurable lesion according to the modified RECIST 1.1 are eligible
4. HER2-low (HER2 1+, HER2 2+ (SISH negative))
5. Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
6. ECOG performance status 0-1 with no deterioration between screening and the first dose of study treatment.
7. Patients must have a life expectancy ≥ 3 months from proposed first dose date.
8. Patients must have had a washout period of 2 weeks for any prior therapy prior to the start of study drug. The following intervals between the end of the prior treatment and first dose of study drug must be observed:

   * Major surgery ≥ 4 weeks
   * Radiation Therapy including palliative stereotactic radiation therapy to chest ≥ 4 weeks
   * Palliative stereotactic radiation therapy to other anatomic areas including whole brain radiation ≥ 2 weeks
   * Anti-Cancer chemotherapy [Immunotherapy (non-antibody based therapy)], retinoid therapy, hormonal therapy ≥ 3 weeks
   * Antibody based anti-cancer therapy ≥ 4 weeks
   * Targeted agents and small molecules ≥ 2 weeks or 5 half-lives, whichever is longer
   * Nitrosoureas or mitomycin C ≥ 6 weeks
   * TKIs approved for treatment of NSCLC ≥1 week (baseline CT scan must be completed after discontinuation of TKI
   * Chloroquine/Hydroxychloroquine ≥ 14 days
   * Cell-free and CART, peritoneal shunt or drainage of pleural effusion, ascites or pericardial effusion ≥ 2 weeks prior to screening assessment
9. Patients must have acceptable bone marrow, liver and renal function measured within 28 days prior to administration of study treatment as defined below:

   * Hemoglobin ≥8.0 g/dL (Red blood cell transfusion is not allowed within 1 week prior to the day)
   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (G-CSF administration is not allowed within 2 weeks prior to the day)
   * Platelet count ≥100 x 109/L (Platelet transfusion is not allowed within 1 week prior to the day)
   * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) or < 3×ULN in the presence of documented Gilbert's syndrome (unconjugated hyperbilirubinemia) or liver metastases at baseline
   * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case it must be ≤ 5x ULN
   * Serum creatinine ≤1.5 x institutional ULN
   * CrCl 30≥mL/min as determined by Cockcroft Gault (using actual body weight)
   * Serum albumin ≥ 2.5 g/dL
   * International normalised ratio or Prothrombin time and either partial thromboplastin or activated partial thromboplastin time ≤ 1.5 × ULN
10. Female patients must be using a highly effective method of contraception (refer to the restrictions on P37) during the clinical trial and for 7 months after permanent discontinuation of the study drug. There must be evidence that patients are not breastfeeding, have a negative pregnancy test, or not of childbearing potential by meeting one of the following criteria at screening:

    1. Post-menopausal women defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatment.
    2. Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but not tubal ligation.
    3. Amenorrhoeic for 12 months and serum follicle-stimulating hormone (FSH), lutenizing hormone (LH) and plasma oestradiol levels in the postmenopausal range for the institution More detailed information is provided in Appendix F (Definition and accepted contraception for women of childbearing age).
11. Non-sterilized male patients who are sexually active with a female partner of childbearing potential must use a condom with spermicide from screening to 4 months after the final dose of IMP. Complete heterosexual abstinence for the duration of the study and drug washout period is an acceptable contraceptive method if it is in line with the patient's usual lifestyle (consideration must be made to the duration of the clinical trial); however, periodic or occasional abstinence, the rhythm method, and the withdrawal method are not acceptable. It is strongly recommended for the female partners of a male patient to also use at least one highly effective method of contraception throughout this period. In addition, male patients should refrain from fathering a child, or freezing or donating sperm from the time of randomisation/enrolment, throughout the study and for 4 months after the last dose of IMP. Preservation of sperm should be considered prior to enrollment in this study.
12. Mandatory biopsy during the screening window prior to dosing and at progression

Exclusion Criteria:

1. Medical history of myocardial infarction within 6 months before registration, symptomatic congestive heart failure (CHF) (New York Heart Association Class II to IV, Section 17.4), troponin levels consistent with myocardial infarction as defined according to American College of Cardiology (ACC) guidelines, unstable angina, or serious cardiac arrhythmia requiring treatment.
2. History of (non-infectious) ILD / pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
3. Has a pleural effusion, ascites or pericardial effusion that requires drainage, peritoneal shunt, or Cell-free and Concentrated Ascites Reinfusion Therapy (CART). (Drainage and CART are not allowed within 2 weeks prior to screening assessment)
4. Has uncontrolled infection requiring IV injection of antibiotics, antivirals, or antifungals.
5. Active hepatitis B or C infection, such as those with serologic evidence of viral infection within 28 days of Cycle 1 Day 1. Subjects with past or resolved hepatitis B virus (HBV) infection who are anti-HBc positive (+) are eligible only if they are HBsAg negative (-). Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
6. Has clinically active brain metastases, defined as untreated and symptomatic, or requiring therapy with steroids or anticonvulsants to control associated symptoms. Subjects with treated brain metastases that are no longer symptomatic and who do not require treatment with steroids for at least three weeks may be included in the study if they have recovered from the acute toxic effect of radiotherapy. A minimum of 2 weeks must have elapsed between the end of whole brain radiotherapy and study enrollment/randomization.
7. Has clinically significant corneal disease in the opinion of the investigator.
8. Prior treatment with an ADC which consists of an exatecan derivative that is a topoisomerase I inhibitor.

   Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than chronic toxicities per the discretion of the investigator, eg, alopecia, peripheral neuropathy, proteinuria, controllable hypertension, and controllable diabetes) not yet resolved to National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0, Grade ≤1 or baseline. Subjects may be enrolled with chronic, stable Grade 2 toxicities (defined as no worsening to >Grade 2 for at least 3 months prior to [randomization/enrollment/Cycle 1 Day 1] and managed with standard of care treatment) that the investigator deems related to previous anticancer therapy, such as:
   * Chemotherapy-induced neuropathy
   * Fatigue
   * Residual toxicities from prior IO treatment: Grade 1 or Grade 2 endocrinopathies which may include:

     1. Hypothyroidism/hyperthyroidism
     2. Type 1 diabetes
     3. Hyperglycaemia
     4. Adrenal insufficiency
     5. Adrenalitis
     6. Skin hypopigmentation (vitiligo)
9. Any gastrointestinal condition that would preclude adequate absorption of afatinib including but not limited to inability to swallow oral medication, refractory nausea and vomiting, chronic gastrointestinal diseases or previous significant bowel resection, intestinal obstruction or CTCAE grade 3 or grade 4 upper GI bleeding within 4 weeks before the enrollment.
10. Active or prior documented autoimmune or inflammatory disorders (including IBD [e.g. Chohn's disease, ulcerative colitis or diverticulitis], SLE, sarcoidosis syndrome, tuberculosis, Wegener syndrome, myasthenia gravis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, at screening. Adjust wording as necessary and consider evaluating at screening for studies with known hepatotoxicity or other relevant requirements, history of organ transplant that requires use of immunosuppressives, glomerulonephritis, nephritic syndrome, Fanconi Syndrome or renal tubular acidosis within the past 2 years prior to the start of treatment. The following are exceptions to this criterion:

    * Subjects with vitiligo or alopecia, hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement or psoriasis not requiring systemic treatment; patients with coeliac disease controlled by diet alone and patients without active disease in the last 5 years may be included after consultation with Chief Investigator.
    * HbsAg carrier without active viral infection and under entecavir prophylaxis will be allowed.
11. Known to have tested positive for human immunodeficiency virus (HIV) (positive HIV 1/2 antibodies) or active tuberculosis infection (clinical evaluation that may include clinical history, physical examination and radiographic findings, or tuberculosis testing in line with local practice). Active or prior documented history of primary immunodeficiency or HIV infection, at screening.
12. Untreated central nervous system (CNS) metastatic disease, leptomeningeal disease, or cord compression. Note: Subjects previously treated for CNS metastases that are asymptomatic, radiographically and neurologically stable for at least 4 weeks and do not require corticosteroids (of any dose) for symptomatic management for at least 4 weeks prior to the first dose of treatment are not excluded.
13. Patients with second primary cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for ≤3 years.
14. Patient was in receipt of any live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving study therapy.
15. Patients currently receiving (or unable to stop use at least 2 weeks) prior to receiving the first dose of afatinib, medications known to be potent inhibitors of CYP1A2 or strong inducers of CYP3A4 with a narrow therapeutic range
16. Patient with any of the following cardiac criteria:

    * Mean QT interval corrected for heart rate (QTc) ≥ 470 ms calculated from electrogram (ECG) using Friderecia's correction
    * Any clinicallly important abnormalities in rhythm, conduction or morphology of resting ECG e.g. complete left bundle branch block, third degree heart block, second degree heart block, PR Interval >250 msec.
    * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, uncorrectable chronic hypokalaemia, congenital long QT syndrome, family history (first-degree relatives) of long QT syndrome or unexplained sudden death under 40 years of age or concomitant medication known to prolong the QT interval
    * Uncontrolled hypotension: systolic BP < 90 mmHg and/or diastolic BP 60 mmHg or clinically relevant orthostatic hypotension, including a fall in blood pressure of > 20 mmHg
    * Atrial fibrillation with a ventricular rate >100 bpm on ECG at rest
    * Symptomatic heart failure (NYHA grade II-IV)
    * Known reduced LVEF < 55%
    * Prior or current cardiomyopathy
    * Prior or current acute myocardial infarction
    * Severe valvular heart disease
    * Uncontrolled angina (Canadian Cardiovascular Society grade II-IV despite medical therapy)
    * Stroke or transient ischaemic attack in prior to screening
    * Acute coronary syndrome within 6 months prior to starting treatment
17. Any evidence of severe or uncontrolled systemic disease, including active infection (requiring antibiotics, antifungals or antivirals), diabetes type I and II, uncontrolled seizures, bleeding diatheses, severe COPD, severe Parkinson's disease.
18. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.

    For unresolved toxicity, A.Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the PI.

    B.Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with Trastuzumab deruxtecan may be included only after consultation with the PI
19. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
20. History of active primary immunodeficiency
21. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 7 months after the last dose of Trastuzumab deruxtecan and Afatinib.
22. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
23. History of allogenic organ transplantation.
24. Lung criteria:

    * Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (e.g. pulmonary emboli within three months of the study enrollment, severe asthma, severe COPD, restrictive lung disease, pleural effusion etc.)
    * Any autoimmune, connective tissue or inflammatory disorders (e.g. Rheumatoid arthritis, Sjogren's, sarcoidosis etc.) where there is documented, or a suspicion of pulmonary involvement at the time of screening. Full details of the disorder should be recorded in the CRF for patients who are included in the study.
    * Prior pneumonectomy (complete)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events by NCI-CTCAE v5.0 | through study completion, an average of 30 months
  Safety and tolerability
ORR (Objective response rate) | through study completion, an average of 30 months
  modified Recist v1.1

SECONDARY OUTCOMES:
Disease Control rate (CR+PR+SD) | through study completion, an average of 30 months
  modified Recist v1.1
Overall survival (OS) | through study completion, an average of 30 months
  Kaplan-Meier method,
Progression free survival (PFS) | through study completion, an average of 30 months
  Kaplan-Meier method,

CONTACTS AND LOCATIONS:
Overall Officials: Jeeyun Lee, Ph, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea